CLINICAL TRIAL: NCT00456794
Title: A 12-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study of the Efficacy of Doses of 20 and 60 mg/Day Istradefylline as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa/Carbidopa
Brief Title: 12-Week, Double-Blind, Placebo-Controlled Study of 20 and 60 mg/Day Istradefylline in Parkinson's Disease Patients on Levodopa/Carbodopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-US-006
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Levodopa; End of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
A 12-week, multicenter, double-blind, randomized study designed to evaluate the safety and efficacy of 20 and 60 mg/day istradefylline compared with placebo in subjects with OFF-time phenomena and advanced Parkinson's disease treated with levodopa/carbidopa.

ELIGIBILITY:
Inclusion Criteria:

1. United Kingdom Parkinson's Disease Society brain bank diagnostic criteria (Steps 1 and 2).
2. Modified Hoehn and Yahr in the OFF state of II-IV.
3. Treated with levodopa/carbidopa for at least one year with a stable regimen for 4 weeks prior to randomization.
4. Taking at least 4 doses of levodopa/carbidopa per day (3 doses if at least 2 doses contained slow-release formulation) with predictable end of dose wearing off.
5. Successfully competed Parkinson's disease patient diary training with at least 120 minutes of OFF time per day.
6. Stable regimen of other antiparkinson's medications for 4 weeks prior to randomization.
7. At least 30 years of age and able to give written informed consent.

Exclusion Criteria:

1. Treatment with liquid levodopa/carbidopa within 4 weeks of randomization.
2. Treatment with MAO inhibitors except selegiline.
3. Treatment within 3 months with centrally acting dopamine antagonists (6 months for depot formulations), e.g., antipsychotic neuroleptics, metoclopramide, buspirone, amoxapine.
4. Neurosurgical operation for Parkinson's disease.
5. Atypical parkinsonism or secondary parkinsonism variants.
6. Diagnosis of cancer or evidence of continued disease within 5 years.
7. Clinically significant illness of any organ system (e.g., ALT or AST > 1.5 times the upper limit of normal).
8. Mini-Mental Status Examination score of 25 or less.
9. History of drug or alcohol abuse or dependence within 2 years.
10. History of psychotic illness or seizures.
11. Clinically relevant depression disorder.
12. History of neuroleptic malignant syndrome.
13. Pregnancy or lactation. Women of child bearing potential must use a reliable method of contraception.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325
Dates: Start 2002-03; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Endpoint in percentage of awake time per day in an OFF state based on the subjects' valid ON/OFF Parkinson's disease diary data.

SECONDARY OUTCOMES:
Actual values and mean change from Baseline in percentage and total hours of awake time per day in the OFF state and ON state, UPDRS I-IV, II and III Scores during ON and OFF states, Global Clinical Impression-Improvement (CGI-I), safety

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sussman, MD, Study Director — Kyowa Kirin, Inc.
Locations (1):
- Contact Kyowa Pharmaceutical, Inc., Princeton, New Jersey, United States

REFERENCES:
- [Derived] Stacy M, Silver D, Mendis T, Sutton J, Mori A, Chaikin P, Sussman NM. A 12-week, placebo-controlled study (6002-US-006) of istradefylline in Parkinson disease. Neurology. 2008 Jun 3;70(23):2233-40. doi: 10.1212/01.wnl.0000313834.22171.17. PMID 18519872